CLINICAL TRIAL: NCT01780831
Title: A Phase I Trial to Evaluate the Safety and Pharmacokinetics of Raltegravir in HIV-1-Exposed Neonates at Risk of Acquiring HIV-1 Infection
Brief Title: Safety and Pharmacokinetics of Raltegravir in HIV-1-Exposed Newborn Infants at Risk of Acquiring HIV-1 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1110; 11891 (Registry Identifier: DAIDS ES); IMPAACT P1110
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): HIV-1-exposed full-term infants. Infants received two single doses of RAL: first dose within 48 hours of birth and second dose at 7-10 days of life:
  * RAL-naive: 3 or 2 mg/kg within 48 hours of birth and 3 mg/kg at 7-10 days of life.
  * RAL-exposed: 1.5 mg/kg within 48 hours of birth and 3 mg/kg at 7-10 days of life.
  Interventions: Drug: Raltegravir
- Cohort 2 (Experimental): HIV-1-exposed full-term infants. Daily RAL through 6 weeks of life with first dosing within 48 hours of birth and between 12-60 hours of birth for in utero RAL-naive and RAL-exposed infants, respectively.
  Daily RAL through 6 weeks of life: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — RAL was given as oral granules for suspension.
  Other Names: ISENTRESS

SUMMARY:
The purpose of this study was to evaluate the safety and pharmacokinetics (PK) of raltegravir (RAL) when given to HIV-1-exposed, normal birth weight newborn infants at risk of acquiring HIV-1 infection. (PK is the study of the time course of absorption, distribution, metabolism, and excretion of drugs in the body.) The primary goal of this study was to determine a dose of RAL that was safe and met the PK targets for infants when administered during the first 6 weeks of life in addition to standard of care antiretroviral (ARV) agents for prevention of perinatal transmission.

DETAILED DESCRIPTION:
This is a Phase I multi-center, open label, non-comparative study to evaluate the safety and PK of RAL administered to HIV-1-exposed full-term (≥37 weeks of gestation) infants when administered during the first 6 weeks of life in addition to the infants' standard HIV-1 ARV prophylaxis.

IMPAACT P1097 (NCT01828073) demonstrated that RAL crossed the placenta from mother to fetus after maternal dosing during pregnancy and RAL was slowly eliminated by the newborn after birth. Therefore, for P1110, within each cohort, infants were stratified into the "RAL-naive" or "RAL-exposed" groups depending on infants' in utero exposure to maternal RAL. The study stratification with respect to in utero RAL exposure allowed for adjustment of the initial RAL dosing (i.e. timing and/or dose size).

Study participants were enrolled in two sequential cohorts with the following actual dosing of RAL in addition to their local standard of care ARV agents for prevention of perinatal transmission. PK and safety data from Cohort 1 (two single doses) provided information for the starting dosing for Cohort 2 (daily dosing through 6 weeks of life).

Cohort 1: Two single RAL doses: first dose within 48 hours of birth and second dose at 7-10 days of life.

* Cohort 1, RAL-naive: 3 or 2 mg/kg within 48 hours of birth and 3 mg/kg at 7-10 days of life. (P1110 V1.0 Clarification Memorandum #3, dated January 15, 2015, adjusted the first dose from 3 mg/kg to 2 mg/kg based on available PK data.)
* Cohort 1, RAL-exposed: 1.5 mg/kg within 48 hours of birth and 3 mg/kg at 7-10 days of life.

Cohort 2: Daily RAL dosing through 6 weeks of life.

* Cohort 2, RAL-naive: Daily dosing through 6 weeks of life with initial RAL dosing within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
* Cohort 2, RAL-exposed: Daily dosing through 6 weeks of life with initial RAL dosing between 12-60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.

Target enrollment was approximately 50 infants and their mothers in order to have a minimum of 12 and 20 PK evaluable infants in Cohorts 1 and 2, respectively. Cohort 1 and Cohort 2 RAL-naive infants (and their mothers) were enrolled under protocol Version 1.0. Cohort 2 RAL-exposed infants (and their mothers) were enrolled under protocol Version 2.0.

Infants and their mothers were enrolled within 48 and within 60 hours of delivery under protocol Versions 1.0 and 2.0, respectively. Infants were followed through 24 weeks of life and their mothers were followed until discharge from the labor and delivery unit.

Infant PK samples were collected as follows:

Cohort 1:

* Dose #1 (within 48 hours of birth) intensive PK sampling: Within 30 min pre-dose, and 1-2 hours post-dose, 4-8 hours post-dose, 12 (±1) hours post-dose, and 24 (±1) hours post-dose.
* One random PK sample at 3-4 days of life.
* Dose #2 (7-10 days of life) limited PK sampling: Within 30 min pre-dose, and 1-2 hours post-dose and 24 (±1) hours post-dose.

Cohort 2:

* Initial dose (within 48 and 12-60 hours of birth for RAL-naive and RAL-exposed infants, respectively) intensive PK sampling: Within 1 hour pre-dose, and 1-2 hours, 6-10 hours, 20-24 hours post-dose.
* PK sampling for second dose: 3-6 hours post-dose.
* PK sampling at 6-9 days of life: Within 1 hour pre-dose of initiating 3mg/kg twice daily.
* Intensive PK sampling at 15-18 days of life: Within 1 hour pre-dose, and 1-2 hours post-dose, 4-6 hours post-dose, and 8-12 hours post-dose.
* PK sampling at 28-32 days of life: Within 1 hour pre-dose of initiating 6 mg/kg twice daily.
* PK sampling at 33-42 days of life done at Week 5-6 visit: Within 1 hour pre-dose, and 3-6 hours post-dose.

Protocol defined infant safety evaluations were done at:

Cohort 1: Entry, 3-4 days of life, 7-10 days of life, 2 weeks of life, 6 weeks of life and 24 weeks of life.

Cohort 2: Entry, 2-4 days of life, 6-9 days of life, 15-18 days of life, 28-32 days of life, 5-6 weeks of life, 8-10 weeks of life and 24 weeks of life.

Infant safety data included death, signs/symptoms, diagnoses and laboratory test results. Laboratory test results included results from evaluations specified in the protocol and evaluations done as part of the infant's clinical care which the sites considered relevant.

PK evaluable infants were those determined by the protocol pharmacologist to have PK results which provide analyzable data on the primary PK parameters of interest. Infants who were PK unevaluable were replaced for PK analysis but continued with the study safety follow-up visits.

Infants were evaluable for safety analysis if they received at least one dose of RAL. The safety analyses were based on data from all safety evaluable infants, regardless of whether they were evaluable for PK analysis.

The study initially opened accrual to Cohort 1 RAL-naive group. The PK and safety data from IMPAACT P1110 Cohort 1 RAL-naive group and from IMPAACT P1097 were used to determine the starting dose for the Cohort 1 RAL-exposed group. Opening accrual to the Cohort 2 RAL-naive group was contingent upon infants enrolled in Cohort 1 RAL-naive and RAL-exposed groups successfully meeting safety criteria and providing adequate PK data to determine a regimen to be tested for daily dosing through 6 weeks of life for the Cohort 2 RAL-naive group. The initial dosing regimen for the Cohort 2 RAL-naive group was determined using population PK modeling and simulations incorporating IMPAACT P1110 Cohort 1 data, along with data from the following IMPAACT studies: P1097, P1066 (NCT00485264) (Cohorts IV and V) and P1026s (NCT00042289). Since the PK results of Cohort 1 RAL-naive and exposed groups were similar except in the first 1-2 days of life and P1097 Cohort 1 results suggested that maternal RAL readily crosses the placenta and results to washout RAL exposure in neonates, Cohort 2 RAL-exposed group was determined to receive the same dose of RAL as Cohort 2 RAL-naive group, except the initial dose for RAL-exposed was delayed to within 12 to 60 hours of life.

ELIGIBILITY:
Maternal Inclusion Criteria:

* Mother is living with HIV and either i) known to have HIV diagnosis prior to labor (testing obtained and designated per local SOC in the medical record and either on or recently started CART prior to delivery) or ii) identified as having HIV diagnosis at the time of labor or in the immediate postpartum period. More information on this criterion can be found in the protocol.
* Risk of mothers transmitting HIV to their infants:

  * Cohort 1 and Cohort 2 (RAL-naive): Mother living with HIV is at "high risk" of transmitting HIV to infant as evidenced by any of the following: Mother has not received any ARV therapy during the current pregnancy prior to the onset of labor and delivery; HIV RNA level greater than 1000 copies/mL within 4 weeks (28 days) prior to delivery; receipt of ARV for less than 4 weeks (28 days) before delivery; on ARVs for 4 weeks or longer but has not taken any ARV for more than 7 days prior to delivery; or mother has documented drug resistant virus to at least one class of ARV drugs.
  * Cohort 2 RAL-exposed: there was no requirement that the mother living with HIV is at "high-risk" of transmitting HIV to her infant.
* Maternal written informed consent for study participation

Maternal Exclusion Criteria:

* Known maternal-fetal blood group incompatibility as evidenced by the presence of an unexpected clinically significant maternal red cell antibody that is known to be capable of causing hemolytic disease of the fetus/newborn
* Mother will be receiving RAL as part of her combination antiretroviral (cART) regimen after delivery and intending to breastfeed her infant
* For Cohort 1 and Cohort 2 RAL-naive groups:

  * Cohort 1 RAL-naive: Mother who received RAL prior to and through delivery unless last RAL dosing during prenatal period was >7 days prior to delivery
  * Cohort 2 RAL-naive: Mother who received RAL prior to and through delivery

Infant Inclusion Criteria:

* Age at enrollment (Note: The full-term infants were HIV-exposed and may have received standard of care ARV prophylaxis/treatment before enrollment):

  * Cohort 1 and Cohort 2 RAL-naive: Aged 48 hours or less.
  * Cohort 2 RAL-exposed: Aged 60 hours or less.
* Infant gestational age at birth at least 37 weeks
* No known severe congenital malformation or other medical condition not compatible with life or that would interfere with study participation or interpretation, as judged by the examining clinician
* Birth weight at least 2 kg
* Able to take oral medications
* Parent or legal guardian able and willing to provide signed informed consent
* For Cohort 1 and Cohort 2 RAL-exposed groups:

  * Cohort 1 RAL-exposed: Infants born to mothers who received RAL during pregnancy with last dose taken within 7 days before delivery.
  * Cohort 2 RAL-exposed: Infants born to a mother who received at least one dose of RAL within 2 to 24 hours prior to delivery.

Infant Exclusion Criteria:

* Infant with bilirubin exceeding the American Academy of Pediatrics guidelines for phototherapy, using the infant's gestational age and risk factors as described in the protocol.
* Clinical evidence of renal disease such as edema, ascites, or encephalopathy.
* Receipt of disallowed medications (phenytoin, phenobarbital, or rifampin).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana F. Clarke, PharmD, Study Chair — Section of Pediatric Infectious Diseases, Boston Medical Center
Locations (15):
- United States (8):
  - Usc La Nichd Crs, Los Angeles, California
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
- Brazil (3):
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan, PR, Puerto Rico
- South Africa (2):
  - Umlazi CRS, Durban, KwaZulu-Natal
  - Fam-Cru Crs, Cape Town
- Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi, Thailand

REFERENCES:
- [Background] Nielsen-Saines K, Watts DH, Veloso VG, Bryson YJ, Joao EC, Pilotto JH, Gray G, Theron G, Santos B, Fonseca R, Kreitchmann R, Pinto J, Mussi-Pinhata MM, Ceriotto M, Machado D, Bethel J, Morgado MG, Dickover R, Camarca M, Mirochnick M, Siberry G, Grinsztejn B, Moreira RI, Bastos FI, Xu J, Moye J, Mofenson LM; NICHD HPTN 040/PACTG 1043 Protocol Team. Three postpartum antiretroviral regimens to prevent intrapartum HIV infection. N Engl J Med. 2012 Jun 21;366(25):2368-79. doi: 10.1056/NEJMoa1108275. PMID 22716975
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, dated December 2004, Clarification August 2009 — https://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 participants were from 2 sites in Brazil, 1 site in South Africa and 7 sites in the USA. Enrollment period was January 2014 - December 2015.
  Cohort 2 participants were from 3 sites in Brazil, 2 sites in South Africa,1 site in Thailand, and 4 sites in the USA. Enrollment period was September 2015 - November 2017.
Groups:
- Cohort 1 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses of RAL: first dose (3 mg/kg or 2mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses of RAL: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 2 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort 2 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 and 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Period: Overall Study
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 2 RAL-naive | Cohort 2 RAL-exposed
Started | 10 | 6 | 26 | 10
Completed | 10 | 6 | 22 | 9
Not Completed | 0 | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled infants.
Groups:
- Cohort 2 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort 2 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL through 6 weeks of life starting between 12 and 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 2 RAL-naive | Cohort 2 RAL-exposed | Total
Number analyzed (Participants) | 10 | 6 | 26 | 10 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 6 | 26 | 10 | 52
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Customized [Median (Full Range); unit: weeks] — Gestational age at birth
  weeks
    Gestational age at birth | 39 [38 to 40] | 38 [37 to 40] | 38 [37 to 41] | 39 [38 to 41] | 39 [37 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 12 | 4 | 24
  Male | 4 | 4 | 14 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 19 | 5 | 30
  Not Hispanic or Latino | 7 | 2 | 7 | 4 | 20
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Birth weight [Median (Full Range); unit: grams] | 3020 [2385 to 4200] | 2948 [2320 to 3385] | 2930 [2390 to 3745] | 3085 [2090 to 4130] | 3000 [2090 to 4200]
Apgar score at 1 minute [Median (Full Range); unit: Scores on a scale] — The APGAR score is an evaluation typically done at 1 minute and 5 minutes after birth to describe an infant's health. It ranges from 0 - 10, where 10 is the best possible score. Baseline table includes Apgar Score at 1 minute after birth.
  Scores on a scale | 8 [8 to 9] | 9 [8 to 9] | 9 [6 to 10] | 9 [8 to 10] | 9 [6 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants Who Died or Had Grade 3/4 Adverse Event Through 6 Weeks of Life
Description: Number of infants who died or had adverse events (AEs) of Grade 3 or 4 as defined in DAIDS AE Grading Table. Events with onset dates prior to first RAL dosing and congenital anomalies assessed as baseline by the study team were considered baseline events and not AEs.
Time Frame: From first dosing of RAL through 6 weeks of life
Population: All infants who received at least one dose of RAL. Excluded one Cohort 2 RAL-naive infant who received one dose of RAL at study entry but was off study right after study entry and thus had no post entry safety data.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses of RAL: first dose (3 mg/kg, 2 mg/kg or 1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 2 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL through 6 weeks of life starting within 48 hours of birth and between 12 to 60 hours of birth for in utero RAL-naive and RAL-exposed infants, respectively: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 1 Total | Cohort 2 RAL-naive | Cohort 2 RAL-exposed | Cohort 2 Total
Number analyzed (Participants) | 10 | 6 | 16 | 25 | 10 | 35
Participants | 2 | 2 | 4 | 7 | 4 | 11
Statistical Analysis 1: Comparison: Cohort 1 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 1 infants who died or had grade 3/4 AE through 6 weeks of life; Clopper-Pearson Confidence Interval (CI) = 25, 90% CI 2-sided [9 to 48.4]
Statistical Analysis 2: Comparison: Cohort 2 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 2 infants who died or had grade 3/4 AE through 6 weeks of life; Clopper-Pearson Confidence Interval (CI) = 31, 90% CI 2-sided [18.7 to 46.6]

2. Primary Outcome: AUC24 for Cohort 1 RAL Dose #1 (Within 48 Hours of Birth)
Description: Area Under the Concentration-time Curve at 24-hour interval (AUC24) based on intensive PK sampling around Cohort 1 RAL dose #1 (within 48 hours of birth)
Time Frame: Cohort 1 RAL dose #1 (within 48 hours of birth) intensive PK sampling: within 30 min pre-dose; and 1-2, 4-8, 12 (±1), 24 (±1) hours post-dose.
Population: All Cohort 1 infants who received the first RAL dosing within 48 hours of birth and had AUC24 data for the dosing. AUC24 was missing for one Cohort 1 RAL-naive infant whose PK samples were possibly switched.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Cohort 1 RAL-naive: 3 mg/kg for First Dose: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (3 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-naive: 2 mg/kg for First Dose: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (2 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-exposed 1.5 mg/kg: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
Arm/Group | Cohort 1 RAL-naive: 3 mg/kg for First Dose | Cohort 1 RAL-naive: 2 mg/kg for First Dose | Cohort 1 RAL-exposed 1.5 mg/kg
Number analyzed (Participants) | 6 | 3 | 6
mg*h/L | 53.88 (34.6) | 44.26 (71.9) | 37.42 (92.7)

3. Primary Outcome: Cmax for Cohort 1 RAL Dose #1 (Within 48 Hours of Birth)
Description: Maximum concentration (Cmax) for Cohort 1 dose #1 (within 48 hours of birth)
Time Frame: Cohort 1 dose #1(within 48 hours of birth) intensive PK sampling: within 30 min pre-dose; and 1-2, 4-8, 12 (±1), 24 (±1) hours post-dose.
Population: All Cohort 1 infants who received the first RAL dosing within 48 hours of birth and had Cmax data for the dosing. Cmax was missing for one Cohort 1 RAL-naive infant whose PK samples were possibly switched.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1 RAL-naive: 3 mg/kg for First Dose: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (3 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-naive: 2 mg/kg for First Dose: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (2 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-exposed: 1.5 mg/kg for First Dose: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
Arm/Group | Cohort 1 RAL-naive: 3 mg/kg for First Dose | Cohort 1 RAL-naive: 2 mg/kg for First Dose | Cohort 1 RAL-exposed: 1.5 mg/kg for First Dose
Number analyzed (Participants) | 6 | 3 | 6
ng/mL | 3360.89 (35.5) | 3405.24 (38.1) | 2188.82 (73.3)

4. Primary Outcome: AUC24 for Cohort 2 Initial RAL Dose (Within 48 and 12-60 Hours of Birth for RAL-naive and RAL-exposed Groups, Respectively)
Description: Area Under the Concentration-time Curve at the 24-hour interval (AUC24) for Cohort 2 initial RAL dose (within 48 and between 12-60 hours of birth for RAL-naive and RAL-exposed, respectively).
Time Frame: Cohort 2 initial dose (within 48 and between 12-60 hours of birth for RAL-naive and RAL-exposed, respectively) intensive PK sampling: within 1 hour pre-dose; and 1-2, 6-10, 20-24 hours post-dose.
Population: All Cohort 2 infants who had AUC24 data for the initial RAL dosing. AUC24 were missing for 2 Cohort 2 RAL-naive infants: one was off-study right after study entry and had incomplete PK specimen collection; and one whose AUC24 could not be estimated due to possible administration of next dose before the 24 hr sample was collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Cohort 2 RAL-naive: 1.5 mg/kg Once Daily on Days 1-7 of Life: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of lifes starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort 2 RAL-exposed: 1.5mg/kg Once Daily on Days 1-7 of Life: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 and 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life
Arm/Group | Cohort 2 RAL-naive: 1.5 mg/kg Once Daily on Days 1-7 of Life | Cohort 2 RAL-exposed: 1.5mg/kg Once Daily on Days 1-7 of Life
Number analyzed (Participants) | 24 | 10
mg*h/L | 38.2 (42) | 42.89 (25.3)

5. Primary Outcome: Clast for Cohort 2 Initial RAL Dose (Within 48 and Between 12-60 Hours of Birth for RAL-naïve and RAL-exposed Groups, Respectively)
Description: Last concentration of the drug (Clast) at 24 hour interval post dosing for the Cohort 2 initial RAL dose (within 48 and at 12-60 hours of birth for RAL-naive and RAL-exposed, respectively). This is the plasma RAL concentration from a sample collected at or close to 24 hours post dose.
Time Frame: Cohort 2 initial dose (within 48 and between 12-60 hours of birth for RAL-naive and RAL-exposed groups, respectively) intensive PK sampling: within 1 hour pre-dose; and 1-2, 6-10, 20-24 hours post-dose.
Population: All Cohort 2 infants who had Clast data for the initial RAL dosing. Clast was missing for one Cohort 2 RAL-naive infant who was off-study right after study entry and had incomplete PK specimen collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 2 RAL-naive: 1.5 mg/kg Once Daily on Days 1-7 of Life: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort 2 RAL-exposed: 1.5 mg/kg Once Daily on Days 1-7 of Life: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 and 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 2 RAL-naive: 1.5 mg/kg Once Daily on Days 1-7 of Life | Cohort 2 RAL-exposed: 1.5 mg/kg Once Daily on Days 1-7 of Life
Number analyzed (Participants) | 25 | 10
ng/mL | 947.90 (84) | 946.24 (74)

6. Primary Outcome: RAL AUC12 for Cohort 2 at 15-18 Days of Life
Description: Area Under the Concentration-time Curve at 12-hour interval (AUC12) of RAL for Cohort 2 at 15-18 days of life.
Time Frame: Intensive PK sampling for Cohort 2 at 15-18 days of life: within 1 hour pre-dose; and 1-2, 4-6, 8-12 hours post-dose.
Population: All infants who continued to receive RAL at or beyond Day 15-18 study visit and had AUC12 for the dosing. AUC12 were missing for 2 RAL-naive infants taken off study prior to Day 15-18 visit; 1 RAL-naive infant with delayed absorption for whom AUC12 could not be estimated; and 1 RAL-exposed infant who had incomplete PK sample collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Cohort 2 RAL-naive: 3 mg/kg Twice Daily on Days 8-18 of Life: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort 2 RAL-exposed: 3 mg/kg Twice Daily on Days 8-28 of Life: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 to 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 2 RAL-naive: 3 mg/kg Twice Daily on Days 8-18 of Life | Cohort 2 RAL-exposed: 3 mg/kg Twice Daily on Days 8-28 of Life
Number analyzed (Participants) | 23 | 9
mg*h/L | 14.3 (49.5) | 18.25 (62.8)

7. Primary Outcome: RAL C12 for Cohort 2 at 15-18 Days of Life
Description: RAL concentration at 12 hours (C12) for Cohort 2 at 15-18 days of life.
Time Frame: Intensive PK sampling for Cohort 2 at 15-18 days of life: within 1 hour pre-dose; and 1-2, 4-6, 8-12 hours post-dose.
Population: All infants who continued to receive RAL at or beyond Day 15-18 study visit and had C12 for the dosing. C12 were missing for 2 RAL-naive infants taken off study prior to Day 15-18 visit; 1 RAL-naive infant with delayed absorption for whom C12 could not be estimated; and 1 RAL-exposed infant who had incomplete PK sample collection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Cohort 2 RAL-naive: 3 mg/kg Twice Daily on Days 8-28 of Life: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 2 RAL-naive: 3 mg/kg Twice Daily on Days 8-28 of Life | Cohort 2 RAL-exposed: 3 mg/kg Twice Daily on Days 8-28 of Life
Number analyzed (Participants) | 23 | 9
mg*h/L | 176.11 (162.1) | 273.59 (176.4)

8. Secondary Outcome: Number of Infants Who Died or Had Grade 3/4 Adverse Event Through 24 Weeks of Life
Description: as for outcome 1
Time Frame: From first RAL dose through 24 weeks of life
Population: All infants who received at least one dose of RAL. Excluded was one Cohort 2 RAL-naive infant who received one dose of RAL at study entry but was off study right after study entry and thus had no post entry safety data.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (3 mg/kg or 2mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single doses: first dose (3 mg/kg, 2 mg/kg or 1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 2 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 to 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life
- Cohort 2 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth and between 12 to 60 hours of birth for in utero RAL-naive and RAL-exposed infants, respectively: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 1 Total | Cohort 2 RAL-naive | Cohort 2 RAL-exposed | Cohort 2 Total
Number analyzed (Participants) | 10 | 6 | 16 | 25 | 10 | 35
Participants | 2 | 2 | 4 | 11 | 4 | 15
Statistical Analysis 1: Comparison: Cohort 1 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 1 infants who died or had grade 3/4 AE through 24 weeks of life; Clopper-Pearson Confidence Interval (CI) = 25, 90% CI 2-sided [9 to 48.4]
Statistical Analysis 2: Comparison: Cohort 2 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 2 infants who died or had grade 3/4 AE through 24 weeks of life; Clopper-Pearson Confidence Interval (CI) = 43, 90% CI 2-sided [28.6 to 58.1]

9. Secondary Outcome: Number of Infants Who Died or Had SADR of Grade 3 or 4 Through 6 Weeks of Life
Description: Number of infants who died or had Suspected Adverse Drug Reaction (SADR) of Grade 3 or 4 as defined in DAIDS AE Grading Table.
  Events with onset dates prior to the first RAL dosing and congenital anomalies assessed as baseline by the study team were considered baseline events and not AEs. SADRs are AEs assessed as definitely related, probably related or possibly related to RAL.
Time Frame: From first RAL dose through 6 weeks of life
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (3 mg/kg or 2mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 1 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (3 mg/kg, 2 mg/kg or 1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort 2 Total: Full term Infants, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth and between 12 to 60 hours of birth for RAL-naive and RAL-exposed infants, respectively: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 1 Total | Cohort 2 RAL-naive | Cohort 2 RAL-exposed | Cohort 2 Total
Number analyzed (Participants) | 10 | 6 | 16 | 25 | 10 | 35
Participants | 1 | 0 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohort 1 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 1 infants who died or had SADR of Grade 3 or 4 through 6 weeks of life; Clopper-Pearson Confidence Interval (CI = 6, 90% CI 2-sided [0.3 to 26.4]
Statistical Analysis 2: Comparison: Cohort 2 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 2 infants who died or had SADR of Grade 3 or 4 through 6 weeks of life; Clopper-Pearson Confidence Interval (CI) = 0 — CI is not provided since the estimation parameter is 0

10. Secondary Outcome: Number of Infants Who Died or Had SADR of Grade 3 or 4 Through 24 Weeks of Life
Description: as for outcome 9
Time Frame: From first RAL dose through 24 weeks of life
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (3 mg/kg or 2 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
Arm/Group | Cohort 1 RAL-naive | Cohort 1 RAL-exposed | Cohort 1 Total | Cohort 2 RAL-naive | Cohort 2 RAL-exposed | Cohort 2 Total
Number analyzed (Participants) | 10 | 6 | 16 | 25 | 10 | 35
Participants | 1 | 0 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohort 1 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 1 infants who died or had SADR of Grade 3 or 4 through 24 weeks of life; Clopper-Pearson Confidence Interval (CI) = 6, 90% CI 2-sided [0.3 to 26.4]
Statistical Analysis 2: Comparison: Cohort 2 Total; Test type: Other — Point and 90% CI estimates of percentage Cohort 2 infants who died or had SADR of Grade 3 or 4 through 24 weeks of life; Clopper-Pearson Confidence Interval (CI) = 0 — CI is not provided since the estimation parameter is 0

11. Secondary Outcome: Cohort 1 Dose #1 Neonatal RAL Elimination (CL/F) by UGT1A1 Genotype Group
Description: Cohort 1 Dose #1 neonatal RAL elimination was represented by Clearance (CL/F), which is the volume of plasma cleared of the drug per unit time. Genotyping for polymorphisms of UGT1A1 were performed on infants who were eligible for PK sampling and were consented by their mothers/guardians (i.e. genotyping was optional) .
Time Frame: Cohort 1 Dose #1 Intensive PK sampling: within 30 min pre-dose; and 1-2, 4-8, 12, 24 hours post-dose. Samples for UGT1A1 genotype testing were collected at study entry.
Population: All Cohort 1 infants with data on CL/F (for dose #1) and UGT1A1 genotype. Excluded were: 1 Cohort 1 RAL-naive infant with missing CL/F due to possible PK specimen switch; 2 Cohort 1 RAL-naive infants with no specimen for genotype testing; 1 Cohort 1 RAL-exposed infant with CL/F and genotype data but was the only infant with (TA)5(TA)6 genotype.
Measure: Median (Inter-Quartile Range); unit: L/hr
Groups:
- (TA)6(TA)6: Cohort 1 infants whose UGT1A1 genotype were (TA)6(TA)6 (wildtype).
- (TA)6(TA)7: Cohort 1 infants whose UGT1A1 genotype were (TA)6(TA)7.
Arm/Group | (TA)6(TA)6 | (TA)6(TA)7
Number analyzed (Participants) | 6 | 6
L/hr | 0.11 [0.10 to 0.13] | 0.06 [0.04 to 0.15]
Statistical Analysis 1: Comparison: (TA)6(TA)6 vs (TA)6(TA)7; Test type: Other; p = 0.298, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Cohort 2 Initial Dose Neonatal RAL Elimination (CL/F) by UGT1A1 Genotype Group
Description: Cohort 2 initial dose neonatal RAL elimination was represented by Clearance (CL/F), which is defined as the volume of plasma cleared of the drug per unit time. Genotyping for polymorphisms of UGT1A1 were performed on infants who were eligible for PK sampling and were consented by their mothers/guardians (i.e. genotyping was optional) .
Time Frame: Intensive PK sampling for Cohort 2 initial dose: within 1 hour pre-dose; and 1-2, 6-10, 20-24 hours post-dose. Samples for UGT1A1 genotype testing were collected at study entry.
Population: All Cohort 2 infants w/ data on initial dose CL/F and UGT1A1 genotype. Exclusions: 1 RAL-naive infant who was off-study right after entry w/ incomplete PK specimens; 1 RAL-naive infant's CL/F can't be estimated due to possible administration of next dose before 24 hr sample collection; 3 RAL-naive and 4 exposed infants w/o genotype specimen.
Measure: Median (Inter-Quartile Range); unit: L/hr
Groups:
- (TA)6(TA)6 Wildtype: Cohort 2 infants whose UGT1A1 genotype were (TA)6(TA)6 (wildtype).
- Mutation: Cohort 2 infants whose UGT1A1 genotype were mutation: (TA)5(TA)5, (TA)5(TA)6, (TA)5(TA)7, (TA)6(TA)7, or (TA)7(TA)7.
Arm/Group | (TA)6(TA)6 Wildtype | Mutation
Number analyzed (Participants) | 15 | 12
L/hr | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
Statistical Analysis 1: Comparison: (TA)6(TA)6 Wildtype vs Mutation; Test type: Other; p = 0.37, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Cohort 2 Neonatal RAL Elimination (CL/F) at 15-18 Days of Life by UGT1A1 Genotype Group
Description: Cohort 2 15-18 days of life dose neonatal RAL elimination was represented by Clearance (CL/F), which is defined as the volume of plasma cleared of the drug per unit time at 15-18 days of life when RAL dosing would have been 3 mg/kg twice daily. Genotyping for polymorphisms of UGT1A1 were performed on infants who were eligible for PK sampling and were consented by their mothers/guardians(i.e. genotyping was optional) .
Time Frame: Intensive PK sampling for Cohort 2 at 15-18 days of life: within 1 hour pre-dose; and 1-2 hours post-dose, 4-6, 8-12 hours post-dose. Samples for UGT1A1 genotype testing were collected at study entry.
Population: All Cohort 2 infants with data on CL/F for Day 15-18 visit & UGT1A1 genotype. Exclusions: 1 RAL-naive infant off-study right after entry w/ incomplete PK specimens; 1 RAL-naive infant withdrew consent; 1 RAL-naive infant stopped RAL after wk 4; 1 RAL-exposed infant w/ incomplete PK specimens; 3 RAL-naive and 4 exposed infants w/o genotype specimen.
Measure: Median (Inter-Quartile Range); unit: L/hr
Arm/Group | (TA)6(TA)6 Wildtype | Mutation
Number analyzed (Participants) | 14 | 11
L/hr | 0.5 [0.4 to 1] | 0.5 [0.4 to 0.8]
Statistical Analysis 1: Comparison: (TA)6(TA)6 Wildtype vs Mutation; Test type: Other; p = 0.98, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Number of Cohort 1 Infants With Hyperbilirubinemia by UGT1A1 Genotype
Description: Hyperbilirubinemia was defined as total bilirubin exceeding 16.0 mg/dL or receipt of phototherapy, or transfusion therapy, or other therapies for hyperbilirubinemia or elevated bilirubin.
Time Frame: Specimens for bilirubin testing were collected at study entry; Days 3-4, 7-10 of life; and Weeks 2, 6, 24 of life for Cohort 1. Specimen for genotype testing was collected at entry.
Population: The intent of this Outcome Measure was to investigate the association between UGT1A1 genotypes with hyperbilirubinemia, however no infants had hyperbilirubinemia.
Groups:
- (TA)5(TA)6: Cohort 1 infants whose UGT1A1 genotype were (TA)5(TA)6.
- (TA)6(TA)7: Cohort 2 infants whose UGT1A1 genotype were (TA)6(TA)7.
Arm/Group | (TA)5(TA)6 | (TA)6(TA)6 | (TA)6(TA)7
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Number of Cohort 2 Infants With Hyperbilirubinemia by UGT1A1 Genotype
Description: as for outcome 14
Time Frame: Specimens for bilirubin testing were collected at study entry; after 2nd dose; Days 6-9, 15-18, 28-32 of life; and Weeks 5-6, 8-10, 24 of life for Cohort 2. Specimen for genotype testing was collected at study entry.
Population: as for outcome 14
Groups:
- (TA)6(TA)6: Cohort 2 infants whose UGT1A1 genotype were (TA)6(TA)6 (wildtype).
- (TA)5(TA)5: Cohort 2 infants whose UGT1A1 genotype were (TA)5(TA)5.
- (TA)5(TA)6: Cohort 2 infants whose UGT1A1 genotype were (TA)5(TA)6.
- (TA)5(TA)7: Cohort 2 infants whose UGT1A1 genotype were (TA)5(TA)7.
- (TA)7(TA)7: Cohort 2 infants whose UGT1A1 genotype were (TA)7(TA)7.
Arm/Group | (TA)6(TA)6 | (TA)5(TA)5 | (TA)5(TA)6 | (TA)5(TA)7 | (TA)6(TA)7 | (TA)7(TA)7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Cohort 1 Infants With Hyperbilirubinemia by SLCO1B3 Genotype
Description: as for outcome 14
Time Frame: Specimens for bilirubin test were collected at study entry; Days 3-4, 7-10 of life; and Weeks 2, 6, 24 of life for Cohort 1. Specimen for genotype testing was collected at study entry.
Population: The intent of this Outcome Measure was to investigate the association between SLCO1B3 genotypes with hyperbilirubinemia, however no infants had hyperbilirubinemia.
Groups:
- C / C: Cohort 1 infants whose SLCO1B3 genotype were C/C (wildtype).
- C / T: Cohort 1 infants whose SLCO1B3 genotype were C/T.
- T / T: Cohorts infants whose SLCO1B3 genotype were T/T.
Arm/Group | C / C | C / T | T / T
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Number of Cohort 2 Infants With Hyperbilirubinemia by SLCO1B3 Genotype
Description: as for outcome 14
Time Frame: as for outcome 15
Population: as for outcome 16
Groups:
- C / C: Cohort 2 infants whose SLCO1B3 genotype was C/C (wildtype).
- C / T: Cohort 2 infants whose SLCO1B3 genotype was C/T.
- T / T: Cohort 2 infants whose SLCO1B3 genotype was T/T.
Arm/Group | C / C | C / T | T / T
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first RAL dose through 24 weeks of life
Description: All Adverse Events (AEs) including diagnoses, signs/symptoms and abnormal laboratory test results mentioned in the "Study Description" section. Events with onset dates prior to first RAL dose and congenital anomalies assessed as baseline by the study team were considered baseline events and not AEs.
Groups:
- Cohort1 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (3 mg/kg or 2 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort1 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: RAL was given as oral granules for suspension. Two single RAL doses: first dose (1.5 mg/kg) within 48 hours of birth and second dose (3 mg/kg) at 7-10 days of life.
- Cohort2 RAL-naive: Full term Infants not exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting within 48 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
- Cohort2 RAL-exposed: Full term Infants exposed in utero to maternal RAL, ≥2000 grams and ≥37 weeks gestational age at birth, born to women living with HIV-1 infection and at risk of acquiring HIV-1 infection.
  Raltegravir: Daily RAL dosing through 6 weeks of life starting between 12 to 60 hours of birth: 1.5 mg/kg once daily during Days 1-7 of life, 3.0 mg/kg twice daily during Days 8-28 of life, and 6.0 mg/kg twice daily during Days 29-42 of life.
Arm/Group | Cohort1 RAL-naive | Cohort1 RAL-exposed | Cohort2 RAL-naive | Cohort2 RAL-exposed
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/25 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/6 | 7/25 | 2/10
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6 | 24/25 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort1 RAL-naive (N=10) | Cohort1 RAL-exposed (N=6) | Cohort2 RAL-naive (N=25) | Cohort2 RAL-exposed (N=10)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Hypertension neonatal (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort1 RAL-naive (N=10) | Cohort1 RAL-exposed (N=6) | Cohort2 RAL-naive (N=25) | Cohort2 RAL-exposed (N=10)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 0
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Laryngomalacia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Pyrexia (General disorders) | 1 | 0 | 7 | 1
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 3 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 8 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 1 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 5 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 4 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 6 | 1
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 4 | 5 | 20 | 7
Neutrophil count decreased (Investigations) | 5 | 4 | 10 | 1
Fontanelle bulging (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | 2
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast induration (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Penile erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 9 | 1
Cyanosis neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5 | 1
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0
Pallor (Vascular disorders) | 0 | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT01780831/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT01780831/SAP_001.pdf